CLINICAL TRIAL: NCT04546451
Title: Musical and Psychomotor Interventions for Cognitive, Sensorimotor, and Cerebral Decline in Patients With Mild Cognitive Impairment (COPE): a Study Protocol for a Multicentric Randomized Controlled Study
Brief Title: Countervail Cognitive and Cerebral Decline in Mild Cognitive Impairment Patients Using Non-medical Interventions
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: University Hospital, Geneva (Other); University of Geneva, Switzerland (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99861
Record Dates: First submitted 2020-08-29; First posted 2020-09-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2022-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Randomized Controlled Trial; Non-medical interventions; Cognitive performance; Sensorimotor performance; Experience induced brain plasticity; Music Practice; Psychomotor training; Passive Control Group; Multivariate data-driven analyses
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: 2 experimental conditions (Music practice vs. Psychomotor training) and 1 passive control condition
Masking Description: Patients will receive the information that 2 interventions to improve cognitive function in Mild Cognitive Impairment will be compared and that assignment to the interventions is random for scientific reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music practice (Experimental): Patients will receive Music Practice interventions of 45 minutes twice a week over 6 months, provided by a professional musician
  Interventions: Behavioral: Music practice
- Psychomotor therapy (Experimental): Patients will receive Psychomotor interventions of 45 minutes twice a week over 6 months, provided by a professional psychomotor therapist
  Interventions: Behavioral: Psychomotor therapy
- Passive control group (No Intervention): Healthy passive controls will pass all measurements without any intervention. The control group participants must adhere to the same inclusion and exclusion criteria as the experimental groups, except for an MCI diagnosis. Control participants will be matched to the experimental groups for age, gender and education level.

INTERVENTIONS:
Behavioral: Music practice — Patients will be trained to play a simple instrument (tongue-drum) in a group setting using different musical styles.
  Arms: Music practice
Behavioral: Psychomotor therapy — Patients will be trained in body awareness and a wide range of of movement activities.
  Arms: Psychomotor therapy

SUMMARY:
Cognitive decline represents a major threat among the deleterious effects of population aging. The investigators propose to conduct an RCT (randomized controlled trial) on the subpopulation of MCI patients, and examine whether intensive musical or psychomotor group interventions can improve their cognitive and sensorimotor functioning, as well as induce brain plasticity, compared to a passive healthy control group, matched for age, gender and education level. The 2 training regimens will take place twice a week over 6 months and will be provided by professionals in each field.

DETAILED DESCRIPTION:
Background Regular cognitive training can boost or maintain cognitive and brain functions known to decline with age. Most studies administered such cognitive training on a computer and in a lab setting. However, everyday life activities, like musical practice or physical exercise that are complex and variable, could be more successful at inducing transfer effects to different cognitive domains and maintaining motivation. "Body-mind exercises", like Tai Chi or psychomotor exercise, may also positively affect cognitive functioning in the elderly. We will investigate the influence of active music practice and psychomotor training over 6 months in Mild Cognitive Impairment patients from university hospital memory clinics on cognitive and sensorimotor performance and brain plasticity.

Methods We aim to conduct a randomized controlled (RCT) multicenter intervention study on 32 Mild Cognitive Impairment (MCI) patients (60-80 years), divided over 2 experimental groups: 1) Music practice; 2) Psychomotor treatment. Controls will consist of a passive test-retest group of 16 age, gender and education level matched healthy volunteers.

The training regimens take place twice a week for 45 minutes over 6 months in small groups, provided by professionals, and patients should exercise daily at home. Data collection takes place at baseline (before the interventions), 3, and 6 months after training onset, on cognitive and sensorimotor capacities, subjective well-being, daily living activities, and via functional and structural neuroimaging. Considering the current constraints of the ongoing COVID-19 (COronaVIrus Disease of 2019) pandemic, recruitment and data collection takes place in 2 waves.

Discussion We will investigate whether musical practice or psychomotor exercise in small groups can improve cognitive, sensorimotor and brain functioning in MCI patients, and therefore provoke benefits for their daily life functioning and well-being.

ELIGIBILITY:
Inclusion criteria

1. MCI diagnosis by experts at the memory clinics
2. MMSE score (Mini-Mental State Examination) > 22 or MoCA (Montreal Cognitive Assessment) > 18
3. Hospital Anxiety and Depression Scale (HADS) < 14 (< 7/21 for anxiety and < 7/21 for depression)
4. Age between 60 and 80 years
5. Right-handedness
6. Fluent in French
7. Able to give informed consent as documented by signature

Exclusion Criteria:

1. Serious motor deficits
2. Impaired/not-corrected hearing
3. Serious physical and mental comorbidities
4. Participation in physical or cognitive training over the last 12 months
5. Maximum 5 years of official music education over the lifespan outside the school curriculum or during the last 3 years
6. Intensive physical activity over the last 12 months (sports or body-mind exercises)
7. Left-handed or ambidextrous
8. MRI incompatibility (claustrophobia, cardiac stimulator, implants…)

Nota bene: for brain organizational reasons exclusively right-handed participants will be included. Right-handed persons represent more than 90% of the population (Isaacs, Barr, Nelson, & Devinsky, 2006., doi:10.1212/01.wnl.0000219623.28769.74.)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
Cognitive Telephone Screening Instrument (COGTEL) | 6 months
  This test can be applied by telephone or face-to-face (in this study we will apply the face-to-face method). The outcome consists of increase or less decrease (experimental group 1 or 2 vs. the control group) of the total weighted score at the COGTEL test directly after the 6 months interventions as compared to directly before the interventions.
  The COGTEL test provides a main weighted score of core cognitive function, it comprises 6 subtests covering prospective memory, short- and long-term verbal memory, working memory (digit span), verbal fluency and inductive reasoning.
  COGTEL main weighted score: COGTEL Total score = 7.2 x Prospective Memory score + 1.0 x Verbal Short-Term Memory score + 0.9 x Verbal Long-Term Memory score + 0.8 x Working Memory score + 0.2 x Verbal Fluency score + 1.7 x Inductive Reasoning score
  (Kliegel, Martin, & Jager, 2007, doi:10.3200/JRLP.141.2.147-172) (lhle et al., 2017, doi:10.1159/000479680)

SECONDARY OUTCOMES:
Individual subtests of the COGTEL (Cognitive Telephone Screening Instrument) | 6 months
  Individual subtests of the COGTEL: prospective memory, short- and long-term verbal memory, working memory (digit span), verbal fluency, and inductive reasoning; the outcome consists of increase or less decrease (experimental group 1 or 2 vs. the control group) of each subtest score directly after the 6 months interventions as compared to directly before the interventions.
D2-R test | 6 months
  D2-R test (attention, processing speed): correct responses/hits minus errors/omissions; the outcome consists of increase or less decrease (experimental group 1 or 2 vs. the control group) of the total score directly after the 6 months interventions as compared to directly before the interventions.
Trail making test | 6 months
  Trail making test A (visual processing speed) & B (visual processing speed & cognitive flexibility): time to complete the test A and B; the outcome consists in decrease or less increase in time to complete the tests (experimental group 1 or 2 vs. the control group) directly after the 6 months interventions as compared to directly before the interventions.
Go/No-Go | 6 months
  Go/No-Go (inhibition): number of errors ; the outcome consists of decrease or less increase (experimental group 1 or 2 vs. the control group) of the total score directly after the 6 months interventions as compared to directly before the interventions.
International Matrix Test (Oldenburg) | 6 months
  Speech-in-noise perception test. The outcome is a score of Speech Reception Threshold (SRT), measured for both ears and each ear separately (Kollmeier et al., 2105, doi: 10.3109/14992027.2015.1020971).
fMRI visual working memory task | 6 months
  fMRI letter n-back visual working memory task (Migo et al., 2015, doi.org/10.1080/13825585.2014.894958): correct responses; the outcome consists of increase or less decrease (experimental group 1 or 2 vs. the control group) of the total score directly after the 6 months interventions as compared to directly before the interventions.
Sensorimotor function | 6 months
  Higher total score of the following sensorimotor tests in the 2 experimental intervention groups as compared to the active control group directly after the 6 months interventions as compared to directly before the interventions.
  1. Clock drawing test (assessing apraxia) (Aprahamian, Martinelli, Neri, & Yassuda, 2009, doi: 10.1590/S1980-57642009DN30200002)
  2. Purdue Pegboard (assessing manual dexterity) (Tiffin & Asher, 1948, doi: 10.1037/h0061266)
  3. Unipedal balance test (Bohannon & Tudini, 2018; doi:10.1016/j.physio.2018.04.001)
  4. Laterality test (assessing left/right judgements) (Williams et al., 2019, doi: 10.1016/j.msksp.2019.01.010)
Short Version of the Amsterdam Instrumental Activity of the Daily Living Questionnaire (A-IADL-Q(SV)) | 6 months
  Daily living activities: improved daily living activities as measured by the A-IADL-Q(SV; Short Version of the Amsterdam Instrumental Activity of the Daily Living Questionnaire) in the 2 experimental intervention groups as compared to the control group directly after the 6 months interventions as compared to directly before the interventions (Jutten et al., 2017, doi:10.1016/j.dadm.2017.03.002).
World Health Organization Quality of Life Instruments - short Version WHOQOL-BREF (abbreviated World Health Organization Quality of Life; WHO 1996) | 6 months
  Subjective well-being: improved subjective well-being in both intervention groups as measured by the WHOQOL-BREF (1996) directly after the 6 months interventions as compared to directly before the interventions. (Organization, W. H. (1996). WHOQOL-BREF: introduction, administration, scoring and generic version of the assessment: field trial version, December 1996.)
Emotional regulation questionnaire (ERQ) | 6 months
  Emotional regulation: improved emotional regulation in the experimental groups as compared to the control group directly after the 6 months interventions as compared to directly before the interventions (Christophe et al., 2009 doi: 10.1016/j.erap.2008.07.001).
Magnetization Prepared 2 Rapid Gradient Echo (MP2RAGE) | 6 months
  MP2RAGE is an extension of the conventional MPRAGE pulse sequence widely used in clinical studies. It involves gray matter volume assessment, allowing to evaluate gray matter changes following learning of new skills (Marques & Gruetter, 2013, doi:10.1371/journal.pone.0069294).
Functional MRI (fMRI) | 6 months
  Letter N-back visual working memory task (Migo et al., 2015, doi.org/10.1080/13825585.2014.894958). Allows evaluating visual working memory performance following learning of new skills.
Resting state functional MRI (RS-fMRI) | 6 months
  RS-fMRI assesses activity in the Default Mode Network (DMN) reflecting global functional connectivity of the brain (Leonardi et al., 2013, doi: 10.1016/j.neuroimage.2013.07.019). Allows evaluating functional connectivity changes following learning of new skills.
Diffusion Tensor Imaging (DTI) | 6 months
  DTI allows computing i.a. Fractional Anisotropy for evaluating white matter integrity reflecting structural connectivity (Bosch et al., 2012, doi: 10.1016/j.neurobiolaging.2010.02.004). Allows evaluating structural connectivity changes following learning of new skills.

CONTACTS AND LOCATIONS:
Overall Officials: Clara E. James, PhD, Principal Investigator — University of Applied Sciences and Arts Western Switzerland, Geneva, Switzerland
Locations (2):
- Switzerland (2):
  - CHUV: Centre Leenaards Memory Center, Lausanne, Canton of Vaud
  - School of Health Sciences Geneva HES-SO, Geneva

IPD SHARING:
Plan to Share IPD: Yes
As soon as the data collection will be completed, all data and all other documents will be stored at YARETA, a FAIR (FAIR data are data which meet principles of findability, accessibility, interoperability, and reusability) digital solution for long-term preservation of research data for all Geneva Universities (https://yareta.unige.ch). The Geneva School of HEalth Sciences already possesses an organizational unit on the YARETA platform.
  The datasets generated during the current study will not publicly available during data collection and analyses. After data collection and analyses completion, they will be published by our research team first, but they will be available in the future from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After study completion (2022)
Access Criteria: To be defined
URL: https://yareta.unige.ch

REFERENCES:
- [Derived] James CE, Stucker C, Junker-Tschopp C, Fernandes AM, Revol A, Mili ID, Kliegel M, Frisoni GB, Brioschi Guevara A, Marie D. Musical and psychomotor interventions for cognitive, sensorimotor, and cerebral decline in patients with Mild Cognitive Impairment (COPE): a study protocol for a multicentric randomized controlled study. BMC Geriatr. 2023 Feb 6;23(1):76. doi: 10.1186/s12877-022-03678-0. PMID 36747142